CLINICAL TRIAL: NCT04331288
Title: PT150 (Formerly ORG34517) as a Potential Treatment for Alcohol Dependence-Alcohol Interaction Study
Brief Title: Effects of Ethanol on the Pharmacokinetics of PT-150 (Formerly ORG34517) (PT150 PK Study)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pop Test Oncology LLC (Industry)
Collaborators: Pharmacotherapies for Alcohol and Substance Use Disorders Alliance (Other); Congressionally Directed Medical Research Programs (U.S. Federal Agency); Michael E. DeBakey VA Medical Center (U.S. Federal Agency); Baylor College of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AS140026-A3c; W81XWH-15-2-0077 (Other Grant/Funding Number: Department of Defense Congressionally Directed Medical Research Program)
Record Dates: First submitted 2020-03-31; First posted 2020-04-02 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-12

CONDITIONS: Potential Treatment for Alcohol Dependence-Alcohol Interaction
Keywords: Alcohol; Alcoholic; Alcoholism; Alcohol abuse; Alcohol interaction; Alcohol Use Disorder; Alcohol use; Alcohol dependence; Alcohol dependent; Post Traumatic Stress Disorder; Substance use Disorder; Ethanol abuse; Ethanol use; Pharmacokinetics
MeSH Terms: conditions — Alcoholism; Alcohol Drinking; Stress Disorders, Post-Traumatic; Substance-Related Disorders | interventions — (11R,13S,17S)-11-(1,3-benzodioxol-5-yl)-17-hydroxy-13-methyl-17-prop-1-ynyl-1,2,6,7,8,11,12,14,15,16-decahydrocyclopenta(a)phenanthren-3-one; Beverages

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PT150 with alcohol consumption (Experimental): Study drug to be administered as a single, fixed dose over a 5-day period. An alcohol challenge will be completed on day 1 (pre-treatment) followed by blood draws over a 24-hour period. PT150 dosing will begin on study day 2 and continue until steady state is reached on day 6, at which point blood draws will occur over a 24-hour period. On day 7, after PT150 steady state has been achieved, an alcohol challenge will be completed followed by blood draws over a 40-hour period.
  Interventions: Drug: PT150; Other: Beverage

INTERVENTIONS:
Drug: PT150 — Intervention 1 includes PT150 with alcohol consumption
  Other Names: Formerly ORG34517
Other: Beverage — The alcohol beverage will be prepared by an in-house pharmacist at the MEDVAMC in a volume of 450 ml for a 70 kg individual and adjusted for body weight by varying the volume. Alcohol will be administered in a concentration of 16% alcohol (Everclear, St. Louis, MO) by volume in juice or another flavored beverage. Participants will be allowed 30 minutes to consume the beverages.
  Other Names: Ethanol beverage

SUMMARY:
The purpose of this clinical study is to assess pharmacokinetic interactions between ethanol (EtOH) and PT150 (900 mg qd) in non-treatment-seeking alcohol-experienced volunteers-(to include military service members, veterans and/or civilians).

DETAILED DESCRIPTION:
This study can be classified as a phase 1, single center, and drug-drug interaction (DDI) study. The within-subjects' experimental procedures will assess pharmacokinetic interactions between ethanol (EtOH) and PT150 (900 mg qd) in non-treatment-seeking alcohol-experienced volunteers (to include military service members, veterans and/or civilians). The specific aim of this study is to evaluate the safety and tolerability of PT150 (a novel, selective Glucocorticoid receptor (GR) antagonist) in combination with alcohol and to determine the amount of PT150 and alcohol in blood (i.e., the pharmacokinetic (PK) interactions between alcohol and PT150) in 10 non-treatment seeking participants. The purpose of this study is to assess the possibility of any adverse interactions between alcohol and PT150. While PT150 might be effective in the treatment of AUD, because alcohol can affect the way that PT150 is metabolized in the body, we first need to determine 1) that it is safe to take PT150 in combination with alcohol, and 2) the amount of PT150 and alcohol in blood after PT150 has reached steady state. This study population will be drawn from adults of any race or ethnicity, males, and females who are post-menopausal, undergoing hormone replacement treatment at a stable dosage for at least 3 months, infertile and not hormone cycling, or using approved non-hormonal contraception for at least two weeks after the last dose. Potential enrollees will be drawn of those NOT seeking treatment for alcohol use disorder (AUD). Statistical goals for the study are to evaluate the pharmacokinetics of PT150 given in combination with exposure to alcohol. The primary objective includes assessing if measures of concentration and timing of PT150 levels in the blood differ between the PT150 challenge (challenge on Day 8 and continually observed through Day 9) in combination with alcohol (ethanol beverage) compared to the steady-state PT150 challenge, absent alcohol challenge, on Day 7. Secondary objectives are to determine if measures of concentration and timing of BAL in the blood differ between the active alcohol challenges only (Day 1/baseline) and PT150 challenges in combination with alcohol challenges (Day 8). Other secondary outcomes include evaluating health and safety outcomes as well as withdrawal from alcohol. After completion of the screening period, the remaining study duration will proceed as follows for each participant: Admission for an initial 1-day in-patient stay; Discharge followed by 4 days of outpatient visits; Readmission for a 4-day inpatient stay; and for females, a follow-up visit will be scheduled to occur at least 14 days after the final dose of PT150 is administered to ensure pregnancy has not occurred. This results in a total participant duration of 10 days.

ELIGIBILITY:
Inclusion Criteria:

1. Provide signed and dated informed consent form;
2. Male or female, aged 21-64;
3. Must score < 10 on the revised clinical institute withdrawal assessment for alcohol scale (CIWA-Ar) assessed in the context of a BAL ≤ 0.00% to demonstrate that they do not need medical detoxification;
4. Must have blood lab test results within the acceptable limits noted in the protocol (Tests may be repeated if initial results are out of range);
5. Have normal vitals (heart rate 50-100 bpm, systolic blood pressure 90-140 mmHg and diastolic blood pressure 60-90 mmHg) and a baseline ECG that demonstrates clinically normal sinus rhythm, clinically normal conduction, normal QTc, and no clinically significant arrhythmias;
6. Have a self-reported medical history and brief physical examination demonstrating no clinically significant contraindications for study participation, in the judgment of the admitting physician;
7. Must be willing to comply with all study procedures and be available for the duration of the study;
8. Women must either be unable to conceive (i.e., surgically sterilized, sterile, or post-menopausal) or using non-hormonal, medically acceptable contraception during the study and for at least 2 weeks after the last dose of study drug has been given, with or without additional hormonal contraception. Women can be receiving hormone replacement treatment (HRT) as long as the HRT dose has been stable for a period of at least 3 months;
9. Women must provide a negative urine pregnancy test within 30 days of alcohol administration on Day 1/baseline (i.e. during the screening period) and a negative serum pregnancy test on day 1 prior to alcohol administration and on day 5. Note that because participants are supervised 24-hours a day when they reside as inpatients, a urine pregnancy test is planned on day 9;
10. Able to provide proof of age and identity (includes providing full name and date of birth).

Exclusion Criteria:

1. DSM-5 criteria for substance use disorders other than alcohol, nicotine, or marijuana or test positive for prescription or illegal substances other than THC. With regard to marijuana/THC, an individual must agree to abstain from marijuana/THC use three days prior to intake (Day 1/baseline);
2. Be pregnant or nursing;
3. Be receiving HRT where their dose has not been stable for a minimum of 3 months;
4. To reduce variability in the magnitude of drug-drug interactions (DDIs), use of concomitant medications (except hormonal birth control) or OTC medications should be excluded for a sufficient time before subject enrollment (at least 14 days or 5 half-lives [whichever is longer]) and for the entire duration of the study. These items should be excluded for a longer time period if the DDI mechanism is induction or time-dependent inhibition. Concomitant medication use includes any prescription, over-the-counter medications or dietary/herbal/nutritional supplements;
5. Be receiving any non-pharmacotherapy treatments or procedures for which there are precautions for taking concomitantly with PT150 and/or those that might interfere with the study;
6. Have neurological or psychiatric disorders other than AUD or SUD for THC;
7. History of suicide attempts and/or current suicidal ideation/plan;
8. Have evidence of untreated or unstable medical illness including: cardiovascular, neuroendocrine, autoimmune, renal, hepatic, or active HIV+, AIDS infection;
9. Have a history of medically adverse reactions to alcohol (e.g., loss of consciousness (LOC), chest pain, or epileptic seizure) or major alcohol-related medical complications requiring hospitalization (i.e. hepatitis or pancreatitis);
10. Have contraindication(s) to take the study medications such as renal or hepatic impairment, congenital metabolic disorders, or hypersensitivity to study medication class (i.e., glucocorticoid antagonists);
11. Have past brain injury/head trauma with current symptoms (e.g. not photophobic, dizziness, etc.) or past report of LOC for >30 minutes and/or have been blast-exposed or had LOC of >1 minute within the last 10 years and current post-concussive symptoms;
12. Self-report more than thirty days' abstinence from alcohol during the three months prior to enrollment/consent;
13. Current signs of violence or aggression assessed as part of the consent process;
14. Participation in a pharmaceutical trial or exposure to investigational drugs within 1 month of the screening visit;
15. Be currently seeking treatment for AUD;
16. Have any other illness, condition, or use medications (psychotropic or antiretroviral), which in the opinion of the PI and/or the admitting physician would preclude safe and/or successful completion of the study;
17. A history of adrenal insufficiency or a baseline plasma cortisol level of ≤ 5mcg/dL;
18. A baseline cortisol of > 5 mcg/dL BUT a post-ACTH stimulation cortisol of <18 mcg/dL;
19. Have been treated with any form of corticosteroid in the past 30 days;
20. Have a history of endometrial hyperplasia, endometrial cancer, uterine polyps, or unexplained vaginal bleeding;
21. Have potassium levels below the normal reference range;
22. Men taking testosterone replacement therapy;
23. Men or women currently interested in fertility;
24. Have underlying inflammatory or auto-immune disorders;
25. Have elevated thyroid stimulating hormone (TSH) levels;
26. Have Type I diabetes.

Ages: 21 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-10-27 (Actual); Study Completion 2023-10-27 (Actual)

PRIMARY OUTCOMES:
Difference in maximum concentration of PT150 (CmaxPT150) | from the PT150 blood draws (days 6-7) to the PT150 with concurrent ethanol blood draws (days 7-9)
  Estimates of maximum concentration (Cmax) of PT150 will be calculated and compared from PT150 steady state alone (days 6-7) to concurrent steady state of PT150 with ethanol exposure (days 7-9).
Difference in time of maximum concentration of PT150 (tmaxPT150) | from the PT150 blood draws (days 6-7) to the PT150 with concurrent ethanol blood draws (days 7-9)
  Estimates of time of maximum concentration (Tmax) of PT150 will be calculated and compared from PT150 steady state alone (days 6-7) to concurrent steady state of PT150 with ethanol exposure (days 7-9).
Difference in terminal elimination half-life of PT150 (t1/2PT150) | from the PT150 blood draws (days 6-7) to the PT150 with concurrent ethanol blood draws (days 7-9)
  Estimates of terminal elimination half-life (T1/2) of PT150 will be calculated and compared from PT150 steady state alone (days 6-7) to concurrent steady state of PT150 with ethanol exposure (days 7-9).
Difference in area under the concentration-time curve of PT150 (AUCPT150) | from the PT150 blood draws (days 6-7) to the PT150 with concurrent ethanol blood draws (days 7-9)
  Estimates of the area under the concentration curve (AUC) through 24 hours post-intervention of PT150 will be calculated and compared from PT150 steady state alone (days 6-7) to concurrent steady state of PT150 with ethanol exposure (days 7-9).

SECONDARY OUTCOMES:
Difference in the maximum concentration of ethanol (CmaxEtOH) | from the ethanol alone blood draws (days 1-2) to the PT150 with concurrent ethanol blood draws (days 7-9)
  Estimates of maximum concentration (Cmax) of ethanol will be calculated and compared from ethanol alone (days 1-2) to concurrent steady state of PT150 with ethanol exposure (days 7-9).
Difference in time of maximum concentration of ethanol (tmaxEtOH) | from the ethanol alone blood draws (days 1-2) to the PT150 with concurrent ethanol blood draws (days 7-9)
  Estimates of time of maximum concentration (Tmax) of ethanol will be calculated and compared from ethanol alone (days 1-2) to concurrent steady state of PT150 with ethanol exposure (days 7-9).
Difference in terminal elimination half-life of ethanol (t1/2EtOH) | from the ethanol alone blood draws (days 1-2) to the PT150 with concurrent ethanol blood draws (days 7-9)
  Estimates of terminal elimination half-life (T1/2) of ethanol will be calculated and compared from ethanol alone (days 1-2) to concurrent steady state of PT150 with ethanol exposure (days 7-9).
Difference in the area under the concentration-time curve of ethanol (AUCEtOH) | from the ethanol alone blood draws (days 1-2) to the PT150 with concurrent ethanol blood draws (days 7-9)
  Estimates of the area under the concentration curve (AUC) through 24 hours post-intervention of ethanol will be calculated and compared from ethanol alone (days 1-2) to concurrent steady state of PT150 with ethanol exposure (days 7-9).
Difference in the number and severity of adverse events | Adverse events are reported throughout the study, from enrollment to study completion
  Difference in the overall number and proportion of adverse events compared among ethanol alone (days 1-2), PT150 alone (days 2-7), and PT150 with ethanol exposure (days 7-9). Comparisons will also be stratified by severity of adverse events.
Difference in heart rate | Heart rate is collected one time after the serial blood draws have been completed for each of ethanol alone (day 2), PT150 alone (day 7), and PT150 with ethanol exposure (day 9).
  Difference in heart rate compared among ethanol alone (days 1-2), PT150 alone (days 6-7), and PT150 with ethanol exposure (days 7-9).
Difference in systolic blood pressure | Systolic blood pressure is collected one time after the serial blood draws have been completed for each of ethanol alone (day 2), PT150 alone (day 7), and PT150 with ethanol exposure (day 9).
  Difference in systolic blood pressure compared among ethanol alone (days 1-2), PT150 alone (days 6-7), and PT150 with ethanol exposure (days 7-9).
Difference in diastolic blood pressure | Diastolic blood pressure is collected one time after the serial blood draws have been completed for each of ethanol alone (day 2), PT150 alone (day 7), and PT150 with ethanol exposure (day 9).
  Difference in diastolic blood pressure compared among ethanol alone (days 1-2), PT150 alone (days 6-7), and PT150 with ethanol exposure (days 7-9).
Change in severity of alcohol withdrawal symptom severity as measured on the Clinical Institute Withdrawal Assessment for Alcohol-Revised (CIWA-Ar) | The CIWA-Ar assessment is completed one time on day 1 prior to ethanol and PT150 exposure, followed by measurements on days 5, 6, 7, 8, and 9 (all post-PT150 exposure measurements).
  Change in CIWA-Ar total score from baseline (pre-PT150 exposure) to all post-PT150 exposure measurements.
Change in ECG abnormalities | An ECG measurement is taken once on day 1 prior to ethanol and PT150 exposure, followed by measurements on days 2, 5, 6, 7, 8, and 9 (all post-PT150 exposure measurements).
  Change in ECG abnormalities from baseline (pre-PT150 exposure) to all post-PT150 exposure measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Verrico, PhD, Principal Investigator — Michael E. DeBakey Veterans Affairs Medical Center
Locations (1):
- Michael E. DeBakey Veterans Affairs Medical Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared with a registry per the data sharing plans of the Consortium